CLINICAL TRIAL: NCT00305604
Title: A Multicenter, Double-Blind, Randomized, Parallel Group Study to Evaluate the Safety and Efficacy of Sitagliptin in Elderly Patients With Type 2 Diabetes Mellitus
Brief Title: Study of Sitagliptin in Older Type 2 Diabetics (0431-047)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-047; MK0431-047; 2006_003
Record Dates: First submitted 2006-03-20; First posted 2006-03-22 (Estimated); Results first posted 2009-05-01 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): sitagliptin
  Interventions: Drug: sitagliptin phosphate
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: sitagliptin phosphate — Once daily (q.d.) administration of sitagliptin 100 mg tablet (or 50 mg based on creatinine clearance). For up to a 24-wk treatment period.
  Other Names: MK0431
  Arms: 1
Drug: Comparator: Placebo — sitagliptin matching placebo for up to a 24-wk treatment period.
  Arms: 2

SUMMARY:
To evaluate the effect of treatment with sitagliptin compared to placebo in elderly patients with type 2 diabetes mellitus who have poor glycemic control with diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling patients 65 years of age or older diagnosed with Type 2 Diabetes not controlled with diet and exercise
* Patients must have a HbA1c of 7-10% off medication, or as a result of a protocol wash-out from oral anti-hyperglycemic agents by the qualifying visit

Exclusion Criteria:

* Patients with type 1 diabetes
* History of ketoacidosis or requires insulin use
* Alanine aminotransferase / aspartate aminotransferase > 2.5 X ULN, triglycerides > 600 mg/dL, creatinine clearance < 35 mL/min
* Fasting plasma glucose consistently > 260 mg/dL
* Poorly controlled hypertension

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 206 (Actual)
Dates: Start 2006-03-08 (Actual); Primary Completion 2008-03-12 (Actual); Study Completion 2008-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Barzilai N, Guo H, Mahoney EM, Caporossi S, Golm GT, Langdon RB, Williams-Herman D, Kaufman KD, Amatruda JM, Goldstein BJ, Steinberg H. Efficacy and tolerability of sitagliptin monotherapy in elderly patients with type 2 diabetes: a randomized, double-blind, placebo-controlled trial. Curr Med Res Opin. 2011 May;27(5):1049-58. doi: 10.1185/03007995.2011.568059. Epub 2011 Mar 23. PMID 21428727

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 30-MAR-2006
  Last Patient Last Visit: 12-MAR-2008
  60 medical clinics in the United States.
Pre-assignment Details: Community dwelling patients ≥ 65 years of age with a diagnosis of type 2 diabetes with hemoglobin A1c (HbA1c) ≥ 7% and ≤ 10% on diet and exercise were eligible to participate. Following a variable duration screening period, patients were randomized in a 1:1 ratio to sitagliptin 100 mg q.d. (or 50 mg q.d. based on creatinine clearance) and placebo.
Groups:
- Sitagliptin: Once-daily administration of sitagliptin 100 mg (or 50 mg based on creatinine clearance); Patients may be down-titrated (1 instead of 2 tablets) if there is a decrease in creatinine clearance to < 50 mL/min at any time during the study.
- Placebo: Sitagliptin-matching placebo tablets.
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 102 | 104
Completed | 70 | 57
Not Completed | 32 | 47
Not completed — Adverse Event | 6 | 3
Not completed — Lack of Efficacy | 11 | 18
Not completed — Lost to Follow-up | 0 | 4
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 12 | 21
Not completed — Patient moved | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 102 | 104 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (6.1) | 72.1 (6.0) | 71.9 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 55 | 109
  Male | 48 | 49 | 97
Race/Ethnicity, Customized [Number; unit: participants]
  White | 76 | 86 | 162
  Black | 10 | 9 | 19
  Hispanic | 9 | 6 | 15
  Asian | 3 | 3 | 6
  Other | 4 | 0 | 4
HbA1c (Hemoglobin A1c) [Mean (Standard Deviation); unit: Percent] | 7.8 (0.8) | 7.8 (0.7) | 7.8 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Hemoglobin A1c) at Week 24
Description: Change from baseline at Week 24 is defined as Week 24 minus Week 0.
Time Frame: Baseline and Week 24
Population: The Full Analysis Set (FAS) included all patients with a baseline value and >= 1 post-baseline value for this outcome. For FAS patients with no data at Week 24, the last observed measurement was carried forward to Week 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 101 | 91
Percent | -0.47 [-0.69 to -0.25] | 0.23 [0.00 to 0.47]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment; baseline; prior anti-hyperglycemic therapy (yes/no); age (< 75/>= 75 yr); baseline creatinine clearance (< 50/>= 50 mL/min); Mean Difference (Net) = -0.70, 95% CI [-0.94 to -0.47], Standard Deviation 0.81

2. Secondary Outcome: Change From Baseline in FPG (Fasting Plasma Glucose) at Week 24
Description: Change from baseline at Week 24 is defined as Week 24 minus Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 96 | 88
mg/dL | -16.2 [-28.9 to -3.6] | 10.6 [-2.7 to 23.9]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -26.8, 95% CI [-40.0 to -13.5], Standard Deviation 45.0

3. Secondary Outcome: Change From Baseline in 2-hour PPG (Post-prandial Glucose) at Week 24
Description: Change from baseline at Week 24 is defined as Week 24 minus Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 74 | 68
mg/dL | -52.1 [-73.6 to -30.7] | 8.9 [-12.4 to 30.1]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -61.0, 95% CI [-82.1 to -40.0], Standard Deviation 63.0

4. Secondary Outcome: Rapidity of Onset of Action as Determined by Home Glucose Monitoring After 1 Week
Description: Fingerstick glucose measurements were taken at 4 times (pre- and 2 hours post-breakfast and dinner) at each of Days -2, 3, and 7. The average of the 4 values was computed for each day. This outcome reflects the Day 7 average minus the Day -2 average.
Time Frame: Week 1
Population: The Full Analysis Set (FAS) included all patients with a baseline value and >= 1 post-baseline value for this outcome. For FAS patients with no data at Day 7, the last observed measurement was carried forward to Day 7. Patients had the option to participate in self monitoring of glucose.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 59 | 62
mg/dL | -25.7 [-34.2 to -17.1] | -2.1 [-10.7 to 6.4]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -23.5, 95% CI [-32.6 to -14.4], Standard Deviation 25.2

ADVERSE EVENTS:
Arm/Group | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 7 | 14
Other Adverse Events (participants affected / at risk) | 4 | 6
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Sitagliptin | Placebo
Any Cardiac disorders (Cardiac disorders) | 1/102 | 4/104
Coronary Artery Disease (Cardiac disorders) | 1/102 | 3/104
Angina Pectoris (Cardiac disorders) | 0/102 | 1/104
Any Gastrointestinal disorders (Gastrointestinal disorders) | 0/102 | 2/104
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0/102 | 1/104
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0/102 | 1/104
Any Hepatobiliary disorders (Hepatobiliary disorders) | 0/102 | 1/104
Cholecystitis (Hepatobiliary disorders) | 0/102 | 1/104
Any Infections and infestations (Infections and infestations) | 3/102 | 3/104
Bronchitis (Infections and infestations) | 1/102 | 0/104
Diverticulitis (Infections and infestations) | 0/102 | 1/104
Mycobacterium Avium Complex Infection (Infections and infestations) | 0/102 | 1/104
Pneumonia (Infections and infestations) | 1/102 | 1/104
Sinusitis (Infections and infestations) | 1/102 | 0/104
Staphylococcal Sepsis (Infections and infestations) | 1/102 | 0/104
Any Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0/102 | 2/104
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0/102 | 1/104
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0/102 | 1/104
Any Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0/102 | 1/104
Dehydration (Metabolism and nutrition disorders) | 0/102 | 1/104
Any Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/102 | 0/104
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/102 | 0/104
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/102 | 0/104
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/102 | 0/104
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/102 | 0/104
Any Renal and urinary disorders (Renal and urinary disorders) | 0/102 | 2/104
Bladder Obstruction (Renal and urinary disorders) | 0/102 | 1/104
Renal Failure Acute (Renal and urinary disorders) | 0/102 | 1/104
Any Reproductive system and breast disorders (Reproductive system and breast disorders) | 0/102 | 1/104
Pelvic Pain (Reproductive system and breast disorders) | 0/102 | 1/104
Any Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0/102 | 1/104
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/102 | 1/104
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Sitagliptin | Placebo
Any Infections and Infestations (Infections and infestations) | 4/102 | 6/104
Urinary Tract Infection (Infections and infestations) | 4/102 | 6/104

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.